CLINICAL TRIAL: NCT04906577
Title: Effects of the Odour of the Very Preterm Infant on Maternal Psychobiology
Acronym: PREMOLF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of logistical problems
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 19-PP-05
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth | interventions — Photography

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VIZOLF (Experimental): visual stimulus (photograph of the child) and olfactory stimulus ad libitum, with a minimum of 6 stimulations per day, to the body odour emitted by the child during the first 5 days of life
  Interventions: Other: photography+odour
- VIZ (Experimental): visual stimulus (photograph of the child) and olfactory stimulus ad libitum, with a minimum of 6 stimulations per day, to a neutral odour during the first 5 days of life
  Interventions: Other: photography

INTERVENTIONS:
Other: photography+odour — Daily from D0 to D5: a square of cotton cloth will be placed against the child's scalp by the childcare worker in charge of the child, then removed and placed in a sealed box containing a photograph of the child, which will then be given to the mother.
  Arms: VIZOLF
Other: photography — A neutral smelling cloth will be placed with the child's photograph which will then be given to the mother.
  Arms: VIZ

SUMMARY:
At birth, the study of interactions, particularly sensory interactions between a mother and her child, allows us to better understand the process of attachment. The sensory signals within the mother-infant dyad will lead to behavioural and metabolic adaptations in both individuals. Currently, the conditions of reception of a very premature newborn in the neonatal intensive care unit of the CHU of Nice lead to a separation between mother and child, with a reduction in sensory interactions.

The immediate and long-term consequences of this "sensory rupture" are widely documented in the child, but little studied in the mother.

The hypothesis at the origin of this work is that olfactory stimulations emanating from the newborn would allow a perceptive continuity between the newborn and his mother. In the pathological situation of the birth of a premature child, these stimulations would lead to neurobiological and behavioural modifications in the mother and would play a role in the attachment process.

ELIGIBILITY:
Inclusion Criteria:

* Immediate postpartum mothers of newborns with a term of < 33 weeks (32 weeks + 6 days)
* primiparous mothers
* Mothers with vaginal delivery, without oxytocin infusion after delivery
* Mothers planning to breastfeed, with no maternal contraindication to breastfeeding

Exclusion Criteria:

* Substance abuse: active smoking at the time of delivery, alcohol, drugs
* Use of medication: antidepressants or psychotropic drugs or centrally acting anti-emetics
* Active depression or history of depression (under medical care with medical follow-up) in the year preceding the birth, on questioning
* Chromosomal abnormality or congenital malformation of pre- or post-natal diagnosis in the newborn
* Language barrier not allowing proper explanation of the protocol and responses to questionnaires

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-09-12 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Change in ocytocine levels | Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Florence CASAGRANDE, Dr, Study Director — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No